CLINICAL TRIAL: NCT06151392
Title: Effect of Probiotic and Zinc Supplementations on the Clinical Outcome in Pediatric Patients with Ventriculitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 195
Record Dates: First submitted 2023-07-22; First posted 2023-11-30 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Ventriculitis, Infectious
Keywords: Probiotic; Zinc; Pediatrics; Ventriculitis
MeSH Terms: conditions — Cerebral Ventriculitis | interventions — Lacteol; Zinc; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Probiotic group (Active Comparator): probiotic will be administered to this group of pediatric patients with ventriculitis
  Interventions: Drug: Probiotic Formula
- Zinc group (Active Comparator): Zinc will be administered to this group of pediatric patients with ventriculitis
  Interventions: Drug: Zinc
- Probiotic and Zinc group (Active Comparator): probiotic and Zinc will be administered to this group of pediatric patients with ventriculitis
  Interventions: Drug: Probiotic Formula; Drug: Zinc
- Control group (No Intervention): interventional drug will not be administered to this group of pediatric patients with ventriculitis

INTERVENTIONS:
Drug: Probiotic Formula — probiotic will be administered to pediatric patients with ventriculitis to study their possible effect in treatment
  Other Names: lactobacillus
  Arms: Probiotic and Zinc group; Probiotic group
Drug: Zinc — Zinc will be administered to pediatric patients with ventriculitis to study their possible effect in treatment
  Other Names: zinc sulfate
  Arms: Probiotic and Zinc group; Zinc group

SUMMARY:
The aim of the study is to evaluate the effect of non-antibiotic-based supplemental interventions in the management of ventriculitis among pediatric patients.

The study objective is to detect the efficacy of probiotics and zinc when taken simultaneously with antibiotic treatment as immunomodulatory in increasing the recovery rate in pediatric population affected with ventriculitis.

DETAILED DESCRIPTION:
Study design: A comparative, randomized, open label, controlled interventional clinical trial.

Setting:The study will be conducted at the Neurosurgery department with the Ain Shams University Hospitals.

Pediatric Patients admitted to the neurosurgery department according to the inclusion criteria will be enrolled in the study and divided into four groups using simple randomization method.

Group A: Patients administer probiotics along with the standard care of therapy for a duration of 14 days.

Lacteol fort ® Sachets manufactured by Rameda contains Lactobacillus LB corresponding to lactobacillus delbruekii and lactobacillus fermentum 10 billion units per sachet.

Dose: 5 billion units once or twice daily. Dosing and duration regimens were guided from Lexicomp Online, Pediatric and Neonatal Lexi-Drugs. https://online.lexi.com. Also, from other studies using probiotics.

Group B: Patients administering zinc supplementation along with the standard care of therapy for the duration of 14 days.

Zn origin® 10 mg/5 mL syrup is manufactured by Egyptian Group for Pharmaceutical Industries. For Origin International Pharma, every 100 mL syrup constituted of 0.8793 g Zn sulfate heptahydrate which contained 0.2 g elemental Zn. Dose:

Infants <3 months: 250 mcg elemental zinc/kg/day. Infants ≥3 months: 100 mcg elemental zinc/kg/day. Dosing and duration regimens were guided from Lexicomp Online, Pediatric and Neonatal Lexi-Drugs. https://online.lexi.com. Also, from other studies using zinc.

Group C: Patients administering probiotics and zinc supplementation along with the standard care of therapy for the duration of 14 days.

Group D: Patients administer only the standard care of therapy (control group). Patient data collection

A. Demographic data:

Including age, sex, weight, height, body mass index.

B. Medication and medical history:

Including patient's medical history, past surgical history, family medical history, and medications the patient is taking or may have recently stopped taking.

A patient's medical history may also include information about allergies, surgeries, immunizations, health habits, such as feeding and sleeping habits.

C. Laboratory examinations The following laboratory data to be measured at baseline and after duration of treatment period of 14 days.

1. CSF culture. Cultures and sensitivity tests from the suspected site of infection were withdrawn from all patients at baseline. Antibiotic susceptibility was carried out using agar diffusion and broth dilution method according to clinical and laboratory standards institute (CLSI) guidelines.
2. CSF chemistry (protein and glucose level). Studies showed that CSF composition comparison had higher leukocyte count in ventriculitis cases. Also, a significantly higher CSF protein and lower CSF glucose value in ventriculitis cases.
3. C-reactive protein (CRP). measured by an immunonephelometric method. CRP is considered an acute phase protein which is synthesized in liver in the presence of infection, it is usually effective in the follow-up of the infection severity.
4. Procalcitonin biomarker. measured by an immunoluminometric assay. It is a 116-amino acid prohormone and is the precursor of hormone calcitonin produced by thyroid gland under normal conditions, the serum concentration of PCT increases significantly during infections. It is secreted from the liver and circulating macrophages in response to infections and could be used for the diagnosis and follow-up.
5. Complete blood picture (CBC) including TLC, RBC, Monocytes and Macrophages.
6. ESR
7. Interleukin-6

D. Signs and symptoms

Follow up the patient signs and symptoms of ventriculitis from hospital admission and during duration of treatment. The Centers for Disease Control and Prevention's National Healthcare Safety Network (CDC/NHSN) definition of healthcare-associated ventriculitis or meningitis includes at least 1 of the following criteria :

Organism cultured from CSF. At least 2 of the following symptoms with no other recognized cause in patients aged >1 year: fever >38°C or headache, meningeal signs, or cranial nerve signs, or at least 2 of the following symptoms with no other recognized cause in patients aged ≤1 year: fever >38°C or hypothermia a <36°C, apnea, bradycardia, or irritability and at least 1 of the following:

* Increased white cells, elevated protein, and decreased glucose in CSF
* Organisms seen on Gram stain of CSF
* Organisms cultured from blood
* Positive nonculture diagnostic laboratory test from CSF, blood, or urine.

E. Safety and Tolerability Evaluation of the safety of probiotic supplementation and zinc in pediatric patients with ventriculitis in terms of side effects and adverse drug events.

F. Patients' follow-up Patients will be followed up during their hospital stay through laboratory examination at baseline and at end of study (14 days).

ELIGIBILITY:
Inclusion Criteria:

• Pediatric patients admitted to neurosurgery department with the diagnosis of ventriculitis will be enrolled in the study.

Exclusion Criteria:

* Patients suffering from any comorbidities other than ventriculitis such as cardiovascular, autoimmune diseases. etc .
* Patients with allergy to zinc.
* Patients with allergy to probiotics.

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CSF culture | after 14 days of treatment
  time-to-event of negative CSF culture .
normalization of the CSF chemistry | after 14 days of treatment
  including normal CSF protein and normal CSF glucose levels
safety of probiotic and zinc supplementation | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events

SECONDARY OUTCOMES:
length of hospital stay | through study completion, an average of 1 year
  number of days the patient stay in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt